CLINICAL TRIAL: NCT01111110
Title: Response to Albuterol Delivered Through an Anti-static Valved Holding Chamber During Nocturnal Bronchospasm
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: Children's Miracle Network (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IRB 103-2008; Children's Miracle Network UFl (Other Grant/Funding Number: Children's Miracle Network, University of Florida)
Record Dates: First submitted 2010-04-23; First posted 2010-04-27 (Estimated); Results first posted 2012-06-19 (Estimated); Last update posted 2022-02-28 (Actual); Status verified 2022-02

CONDITIONS: Asthma
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Anti-static then Static for Albuterol (Experimental): albuterol anti-static first then static chamber second.
  Interventions: Device: anti-static then static
- Static then Anti-static for Albuterol (Experimental): static then antistatic albuterol
  Interventions: Device: Static then anti-static chamber

INTERVENTIONS:
Device: anti-static then static — Albuterol using static chambers
  Arms: Anti-static then Static for Albuterol
Device: Static then anti-static chamber — albuterol with Static then anti-static chambers
  Arms: Static then Anti-static for Albuterol

SUMMARY:
Delivery of HFA albuterol through an antistatic valved holding chamber (VHC) will improve bronchodilator response during nocturnal bronchospasm.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-65 years.
* Physician diagnosis of asthma.
* FEV1 60-80% predicted during the day.
* FEV1 increases ≥ 12 % and to ≥ 80% predicted after 2- 4 puffs of albuterol HFA MDI delivered by antistatic VHC.
* No smoking in the previous year and < 10-pack year history.
* No history of severe asthma attacks requiring ER visit or hospitalization in the previous three months.

Exclusion Criteria:

* Patient required a short course of oral steroid in the past 30 days.
* Any disease that is inadequately controlled or any medication that would worsen asthma or interact with asthma medications.
* History of viral respiratory tract infection in the 3 weeks prior to the screening visit.
* Positive pregnancy test.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 88 (Actual)
Dates: Start 2008-05; Primary Completion 2009-04 (Actual); Study Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- University of Florida, Gainesville, Florida, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment process was done in the Asthma Research Lab. Note that 88 were screened and 4 subjects randomized but determined to be ineligile before starting treatment. They are amongst the screen failures.
Pre-assignment Details: Subjects qualified in the screening visit went into a 7 day run-in-period They needed to have a 20% peak flow overnight drop on 3/7 nights in order to qualify for overnight stays in the Clinical Research Center. Arms are identified by order of treatment assignment. Any other designation is not consistent with our protocol requirements.
Groups:
- Anti-static/Static: albuterol with anti-static chamber then Static on another night
- Static/Antistatic: albuterol with static chamber then with antistatic chamber on another night.
Period: Overall Study
Arm/Group | Anti-static/Static | Static/Antistatic
Started | 3 | 4
Completed | 3 | 4
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Anti-static/Static | Static/Antistatic | Total
Number analyzed (Participants) | 3 | 4 | 7
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 3 | 4 | 7
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 28.3 (11.1) | 21.5 (2.8) | 24.4 (7.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 2 | 1 | 3
Region of Enrollment [Number; unit: participants]
  United States | 3 | 4 | 7

OUTCOME MEASURES:

1. Primary Outcome: Y=100([FEV1 at 1 Puffs-FEV1 at 4AM)/FEV1@4AM] Difference Period 2 Minus Period 1.
Description: (Percent improvement in FEV1 (Forced Expiratory Volume and Forced Vital Capacity) Post Dose for Period 2 over 4AM Baseline value) less (Percent improvement in FEV1 Post Dose for Period 1 over 4AM Baseline value) when 1 Puff go into chamber
Time Frame: fifteen minutes after 1 puff of albuterol
Population: Study intended to get more subjects, but PI's review committee had to deal with candidate deadlines and a high rate of screen failures and allowed her to test seven subjects. Primary concern was the research experience, not the study questions. There was no bias in failing to meet accrual objectives thanks to the blinding.
Measure: Mean (Standard Error); unit: percentage of change from 4AM
Arm/Group | Anti-static/Static | Static/Antistatic
Number analyzed (Participants) | 3 | 4
percentage of change from 4AM | -15.4 (12.2) | 26.7 (20.3)
Statistical Analysis 1: Comparison: Anti-static/Static vs Static/Antistatic; (Comparison of period 2 minus period 1) results Point and interval estimates are halved because this estimates twice the effect size; Test type: Superiority or Other; p = 0.026, t-test, 2 sided; two sample effect size must be halved to account for mean difference estimates twice the effect size; half the mean difference = 21.0, 95% CI 2-sided [3.8 to 41.7], Standard Error of Mean 6.7 — See 4 Puff result

2. Primary Outcome: Y=100([FEV1 at 2 Puffs-FEV1 at 4AM)/FEV1@4AM] Difference Period 2 Minus Period 1.
Description: (Percent improvement in FEV1(Forced Expiratory Volume and Forced Vital Capacity) Post Dose for Period 2 over 4AM Baseline value) less (Percent improvement in FEV1 Post Dose for Period 1 over 4AM Baseline value) when 2 Puffs go into chamber
Time Frame: 15 minutes after 2 puffs of albuterol
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change from 4AM
Arm/Group | Anti-static/Static | Static/Antistatic
Number analyzed (Participants) | 3 | 4
percentage of change from 4AM | -15.3 (14.1) | 31.8 (19.8)
Statistical Analysis 1: Comparison: Anti-static/Static vs Static/Antistatic; Study intended to get more subjects, but PI's review committee had to deal with candidate deadlines and a high rate of screen failures and allowed her to test seven subjects. Primary concern was the research experience, not the study questions. There was no bias in failing to meet accrual objectives thanks to the blinding; Test type: Superiority or Other; p = 0.018, t-test, 2 sided — The effect size is half the difference between the means as (A-B)-(B-A)=2A-2B; Must take half the mean difference to estimate effect size; half the mean difference = 23.5, 95% CI 2-sided [6.0 to 41.0], Standard Error of Mean 6.8 — No comments

3. Primary Outcome: Y=100([FEV1 at 4 Puffs-FEV1 at 4AM)/FEV1@4AM] Difference Period 2 Minus Period 1.
Description: (Percent improvement in FEV1 (Forced Expiratory Volume and Forced Vital Capacity) Post Dose for Period 2 over 4AM Baseline value)less (Percent improvement in FEV1 Post Dose for Period 1 over 4AM Baseline value) when 4 Puffs go into chamber
Time Frame: fifteen minutes after 4 puffs of albuterol
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of change from 4AM
Arm/Group | Anti-static/Static | Static/Antistatic
Number analyzed (Participants) | 3 | 4
percentage of change from 4AM | -17.5 (13.6) | 31.9 (19.3)
Statistical Analysis 1: Comparison: Anti-static/Static vs Static/Antistatic; Null hypothesis is that the Treatment order is independent of the dependent variable based on Period 2 minus Period 1; Test type: Superiority or Other; p = 0.013, t-test, 2 sided; Effect size=half the mean diff = 24.7, 95% CI 2-sided [7.7 to 41.7], Standard Error of Mean 6.6 — You kicked this out on another trial, but note that the period 2-Period 1 differences between the orderings estimate twice the effect size. The effect sizes herein take this into account

ADVERSE EVENTS:
Groups:
- Static: albuterol with static chamber
- Antistatic: albuterol with antistatic chamber.
Arm/Group | Static | Antistatic
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/7
Other Adverse Events (participants affected / at risk) | 0/7 | 0/7

LIMITATIONS AND CAVEATS:
Nocturnal asthma model is a very sensitive model, but very labor intensive and to get more completed subjects, we might need to do multicenter trial

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No